CLINICAL TRIAL: NCT01824563
Title: Benefits of the HiResolutionTM Bionic Ear System in Adults With Low-Frequency Hearing.
Status: Completed | Type: Observational
Sponsor: Advanced Bionics AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AB-RCA-01-2013
Record Dates: First submitted 2013-03-22; First posted 2013-04-05 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Severe-to-profound Hearing Loss
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- study population: Subjects will need to be standard CI patients acording to national implant criteria and the study criteria.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study

SUMMARY:
The goal of this investigation is to generate the needed PMCF data for the HiFocus Mid-Scala electrode. As a point of interest the investigators would like to evaluate the benefit to patients with low-frequency residual hearing implanted with the HiFocus Mid-Scala Electrode. The HiFocus Mid-Scala electrode array is designed to allow surgeons the flexibility to use a variety of contemporary surgical techniques that have been shown to enable easy insertion and to minimize cochlear trauma (see, e.g., Adunka and Buchman, 2007; Friedland and Runge-Samuelson, 2009; Roland et al., 2007). Temporal bone experiments have shown the HiFocus Mid-Scala electrode array to be straightforward to insert while causing minimal trauma to cochlear structures during and after surgery (Lenarz et al., 2010). In addition , the HiFocus Mid-Scala has already shown to be a safe electrode and promising post op clinical results in the premarketing study that is now in the final stage.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Definite Postlingual onset of severe-to-profound hearing loss as documented by completing main stream primary education.
* Local language proficiency
* Bilateral, sensorineural hearing loss

Exclusion Criteria:

* Previous inner ear surgery or active middle ear pathology.
* Cochlear malformation or obstruction
* Presence of additional disabilities that would prevent or interfere with participation in the required study procedures
* Medical or psychological conditions that contraindicate surgery or impact the ability to manage an implanted device or the study-related procedures
* Evidence of central auditory lesion or compromised auditory nerve
* Concurrent participation in other study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: individuals with severe-to-profound hearing loss
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
CI aided word recognition scores in quiet and noise. | 12 months post activation
  CI aided word recognition scores in quiet and noise.

OTHER OUTCOMES:
Evaluate the potential of preservation of residual low frequency hearing | 12 months
  Evaluate the difference in Pure tone thresholds pre and post implantation in the low frequencies.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Frijns, Prof Dr, Principal Investigator — LUMC - Department of ORL-HNS
Locations (1):
- Leiden University Medical Centre, Leiden, Netherlands